CLINICAL TRIAL: NCT01687036
Title: Cryoablation of Atrial Fibrillation Using a Novel Cryoablation System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: afreeze GmbH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CoolLoop First
Record Dates: First submitted 2012-07-18; First posted 2012-09-18 (Estimated); Results first posted 2014-01-13 (Estimated); Last update posted 2018-12-06 (Actual); Status verified 2018-11

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Cryoablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cryoablation (Other): Cryoablation
  Interventions: Device: Cryoablation

INTERVENTIONS:
Device: Cryoablation — Cryoablation of Atrial Fibrillation Using a Novel Cryoablation System
  Other Names: Cool Loop first; Cryoablation of Atrial Fibrillation

SUMMARY:
Primary Endpoint Safety and tolerability of ablation using the AFreeze Cryoablation System consisting of the ablation CoolLoop® catheter, its steerable sheath and the cryoconsole Cryo-Caddy will be assessed and expressed in number of participants with Adverse Events (AEs).

DETAILED DESCRIPTION:
Therefore, the primary endpoint will be a measurement of the following parameters and expressed in number of participants with AE:

* deformation of the catheter loop resulting in entrapment of the catheter in the heart and difficulties removing the catheter during visit 3 (treatment)
* phrenic nerve palsy during visit 3 (treatment)- onset and time course between visit 3 (treatment) and visit 5 (discharge) of death, pericardial tamponade, valve damage requiring surgery and hemorrhage requiring transfusion.
* onset and time course between visit 3 (treatment) and visit 9 (final visit) of atrioesophageal fistula, sepsis, abscesses, endocarditis, stroke, transient ischemic attack, and pulmonary vein (PV) stenosis requiring intervention.

Secondary Endpoint

The following parameters will be assessed and expressed in number of participants with AE/duration time:

* feasibility, defined by the ability to position the catheter in the proximal part in each of the PVs using an over-the-wire technique, forming the cryo-applicator of the catheter to a loop by operating the catheter handle, position-ing the loop at the wall of the PV antrum and delivering cryothermia.
* acute efficacy of catheter ablation is defined as the percentage of electrodes within the PV without measureable signals.
* clinical efficacy of catheter ablation defined by freedom of Atrial Fibrillation (AF) four, eight and twelve weeks after ablation.
* procedure time defined from introduction of the CoolLoop® catheter into the left atrium until removal of the CoolLoop® catheter from the left atrium after termination of the last cryoapplication.
* fluoroscopy time defined from introduction of the CoolLoop® catheter into the left atrium until removal of the CoolLoop® catheter from the left atrium after termination of the last cryoapplication.
* cumulative cryoablation time.
* onset and time course between visit 3 (treatment) and visit 5 (discharge) of pneumothorax, hemothorax, femoral pseudoaneurysm, arteriovenous fistulae, hemorrhage not requiring transfusion.

ELIGIBILITY:
Inclusion Criteria:

* age 18 - 70 years
* symptomatic paroxysmal AF, according to the actual guidelines of the Eu-ropean Society of Cardiology, despite treatment with at least one antiarr- hythmic drug
* at least one episode of AF within the last 3 months documented by ECG
* signed and dated informed consent documented by the patient, indicating that the patient has been informed of all the pertinent aspects of the trial prior to study enrollment
* female subjects of childbearing potential can be included, if they: agree to use, and be able to comply with, effective contraception without in-terruption, from study enrollment, throughout hospitalization and until 12 weeks after catheter ablation (day 0, visit 3). This applies unless the subject commits to absolute and continued abstinence. The following are effective methods of contraception:
* Implant,
* Levonorgestrel-releasing intrauterine system (IUS),
* Medroxyprogesterone acetate depot,
* Tubal sterilization,
* Sexual intercourse with a vasectomized male partner only; vasectomy must be confirmed by two negative semen ana-lyses,
* Ovulation inhibitory progesterone-only pills (i.e., desoge-strel). (Combined oral contraceptive pills are not recommended. If a subject was using combined oral contraception, she must switch to one of the methods above. The increased risk of venous thromboembolism (VTE) continues for 4 to 6 weeks after stopping combined oral contraception.

Exclusion Criteria:

* left atrial diameter > 50 mm as assessed by transthoracic echocardiogra-phy,
* electrical cardioversion performed later than seven days after onset of AF,
* advanced structural heart disease including
* moderate-to-severe valvular stenosis or regurgitation,
* previous myocardial infarction with impaired left ventricular systolic function,
* congenital heart disease,
* left ventricular ejection fraction < 45% during sinus rhythm,
* coronary artery bypass graft surgery within the last 3 months.
* chronic obstructive pulmonary disease treated with beta-sympathomimetic drugs,
* severe respiratory insufficiency,
* known bleeding diathesis or intolerance of heparin or oral anticoagulation,
* previous AF ablation,
* left atrial thrombus,
* severe comorbidity,
* hyperthyreosis,
* any condition, including the presence of laboratory abnormalities, which would place the subject at unacceptable risk if he / she were to participate in the study or confound the ability to interpret data from the study,
* any serious medical condition, laboratory abnormality, or psychiatric illness, that would prevent the subject from signing the Informed Consent Form,
* pregnant or lactating females,
* other severe conditions, which makes the patient unsuitable to participate in the study, as judged by the Investigator,
* the patient is active in another clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-09; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Markus Stuehlinger, MD, Principal Investigator — Medical University Innsbruck
Locations (2):
- Austria (2):
  - Medical University Innsbruck, Innsbruck
  - AKH Linz, Linz

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: September 3,2012 - December 14, 2012 Locations: Medical University Innsbruck, General Hospital Linz
Groups:
- Cryoablation: Cryoablation
  Cryoablation : Cryoablation of Atrial Fibrillation Using a Novel Cryoablation System (single treatment during visit 3).
Period: Overall Study
Arm/Group | Cryoablation
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Cryoablation: Cryoablation
  Cryoablation : Cryoablation of Atrial Fibrillation Using a Novel Cryoablation System
Arm/Group | Cryoablation
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Region of Enrollment [Number; unit: participants]
  Austria | 10

OUTCOME MEASURES:

1. Primary Outcome: Safety of Ablation Using the AFreeze Cryoablation System Consisting of the CoolLoop® Ablation Catheter, Its Steerable Sheath and the Cryoconsole Cryo-Caddy Assessed by Recording All Serious Adverse Events (SAEs)
Description: The primary study objective is assessed by recording all Serious Adverse Events (SAEs).
  Primary endpoint: measurement of the following parameters:
  * deformation of the catheter loop resulting in entrapment of the catheter in the heart and difficulties removing the catheter during visit 3 (treatment).
  * phrenic nerve palsy during visit 3 (treatment).
  * onset and time course between visit 3 (treatment) and visit 5 (discharge) of death, pericardial tamponade, valve damage requiring surgery and hemorrhage requiring transfusion.
  * onset and time course between visit 3 (treatment) and visit 9 (final visit) of atrioesophageal fistula, sepsis, abscesses, endocarditis, stroke, transient ischemic attack, and PV stenosis requiring intervention.
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Cryoablation
Number analyzed (Participants) | 10
participants | 6

2. Primary Outcome: Tolerability of Ablation Using the AFreeze Cryoablation System
Description: The primary study objective is assessed by recording all Adverse Events (AEs).
  Primary endpoint: measurement of the following parameters:
  - deformation of the catheter loop resulting in entrapment of the catheter in the heart and difficulties removing the catheter during visit 3 (treatment).
Time Frame: Treatment duration, up to 6 hours
Measure: Number; unit: AE (device related)
Arm/Group | Cryoablation
Number analyzed (Participants) | 10
AE (device related) | 1

3. Secondary Outcome: Feasibility of Catheter Ablation Measured by Number of Participants Treated With the AFreeze Cryoablation System.
Description: Feasibility, defined by the ability to position the catheter in the proximal part in each of the pulmonary veins (PVs) using an over-the-wire technique, forming the cryo-applicator of the catheter to a loop by operating the catheter handle, positioning the loop at the wall of the PV antrum and delivering cryothermia.
Time Frame: Treatment Duration
Measure: Number; unit: participants
Arm/Group | Cryoablation
Number analyzed (Participants) | 10
participants | 10

4. Secondary Outcome: Acute Efficacy of Catheter Ablation
Description: Absolute percentage of PVs isolated with the CoolLoop® catheter.
Time Frame: Treatment Duration
Measure: Number; unit: percentage of isolated PVs
Arm/Group | Cryoablation
Number analyzed (Participants) | 10
percentage of isolated PVs | 57.5

5. Secondary Outcome: Clinical Efficacy of Catheter Ablation
Description: During follow-up recurrence of AF was reported by the patient and documented by ECG in 8 patients (80%). 2 patients remained free of recurrences of AF.
Time Frame: First patient - first visit: September 11, 2012; Last patient - last visit: March 26, 2013
Measure: Number; unit: participants
Arm/Group | Cryoablation
Number analyzed (Participants) | 10
participants | 2

6. Secondary Outcome: Procedure Time
Description: Procedure time was defined from introduction of the CoolLoop® catheter into the left atrium until removal of the CoolLoop® catheter from the left atrium after termination of the last cryo-application.
Time Frame: Average procedure time: 251 min. 06 sec. (range 126 - 320 min.)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Cryoablation
Number analyzed (Participants) | 10
minutes | 251.1 (59.7)

7. Secondary Outcome: Fluoroscopy Time
Description: Fluoroscopy time was defined from introduction of the CoolLoop® catheter into the left atrium until removal of the CoolLoop® catheter from the left atrium after termination of the last cryo - application. Accumulated time using fluoroscopy during procedure time.
  Average fluoroscopy time was 44 min. 01 sec. (range 17 min. 03 sec. - 59 min.).
Time Frame: Treatment Duration
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Cryoablation
Number analyzed (Participants) | 10
minutes | 44 (13.2)

8. Secondary Outcome: Cumulative Cryoablation Time
Description: Cryoablation time was defined as the cumulative duration of all cryoapplications in each single study patient.
  Average cryoablation time was 114 min. 33 sec. (range 80 - 130 min.).
Time Frame: First patient - first visit: September 11, 2012; Last patient - last visit: March 26, 2013
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Cryoablation
Number analyzed (Participants) | 10
minutes | 113.9 (18.1)

9. Secondary Outcome: AE
Description: 18 AEs were recorded in 7 out of 10 patients. 3 AEs were definitely related to treatment and one AE was definitely device related. All patients recovered completely.
Time Frame: First patient - first visit: September 11, 2012; Last patient - last visit: March 26, 2013
Measure: Number; unit: participants
Arm/Group | Cryoablation
Number analyzed (Participants) | 10
participants | 7

ADVERSE EVENTS:
Time Frame: First patient - first visit: September 11, 2012; Last patient - last visit: March 26, 2013 (6 months and 15 days)
Description: Patients were closely followed for adverse events during treatment and within the defined follow up period according to the study protocol. All Adverse Events including intercurrent disease had to be documented in the patient's medical file and subsequently in the case report form.
Arm/Group | Cryoablation
Serious Adverse Events (participants affected / at risk) | 6/10
Other Adverse Events (participants affected / at risk) | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cryoablation (N=10)
groin hematoma (Surgical and medical procedures) | 1 (1) — Groin hematoma with arterial bleeding from arteria femoralis sin. during puncture of vena femoralis sin. Bleeding stopped by surgical Intervention.
Hospitalization (Cardiac disorders) | 5 (5) — Hospitalization due to recurrent atrial fibrillation.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cryoablation (N=10)
air embolism (Vascular disorders) | 1 (1) — air embolism (after introduction of investigational device into left atrium ST-Elevation in ECG observed; transient Hypotension)
neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) — neck pain (Mb. Bechterew)
hyperthyreosis factitis (Endocrine disorders) | 1 (1)
groin hematoma with art. bleeding (Vascular disorders) | 1 (1)
anemia (Blood and lymphatic system disorders) | 1 (1) — anemia due to art. bleeding
back pain (Musculoskeletal and connective tissue disorders) | 3 (3) — back pain
atrial fibrillation (Cardiac disorders) | 2 (2) — recurrent atrial fibrillation
Hospitalization (Cardiac disorders) | 2 (2) — Hospitalization due to recurrent atrial fibrillation
catheter loop not retractable to straight position (Surgical and medical procedures) | 1 (1) — Catheter loop not retractable to straight position; catheter could be retracted after "rescue maneuver" as defined in the system's user manual.
dyspepsia (Gastrointestinal disorders) | 1 (1)
burning eyes (Eye disorders) | 1 (1)
dyscardia (Cardiac disorders) | 1 (1)
intermittent ST elevation (Vascular disorders) | 1 (1) — intermittent ST elevation (susp. air embolism). ST elevation: finding on an electrocardiogram, wherein the trace in the ST segment is abnormally high above the isoelectric line.
dizzyness (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following approval of the Sponsor and before publishing or presenting data related to the Trial or the Device, Research lnstitution, Principal lnvestigator, and Co-lnvestigator agree to submit copies of any and all proposed manuscripts or abstracts to Sponsor at least 30 days in advance of the date that the applicable party proposes to submit such proposed manuscripts or abstracts to a publisher or other third party.